CLINICAL TRIAL: NCT04226885
Title: Comparison of Nebulized Fentanyl, Midazolam and Dexmedetomidine as a Sedative Premedication in Outpatient Pediatric Dental Surgeries : A Randomized Double Blind Study.
Brief Title: Comparison of Nebulized Fentanyl, Midazolam and Dexmedetomidine as a Premedication in Pediatric Dental Surgeries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Marwa Mohamed Medhat, lecture of anesthesia and surgical intensive care, Zagazig University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 5742-3-12-2019
Record Dates: First submitted 2020-01-05; First posted 2020-01-13 (Actual); Last update posted 2021-04-21 (Actual); Status verified 2021-04

CONDITIONS: Dental Surgeries
Keywords: fentanyl ,midazolam, dexmeditomidine
MeSH Terms: interventions — Fentanyl; Midazolam; Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- fentanyl (Active Comparator): patients will be given nebulized fentanyl 2μg/kg body weight 30 min before surgery
  Interventions: Drug: fentanyl
- midazolam (Active Comparator): The patients will be given nebulized midazolam 0.2 mg/kg body weight 30 min before surgery.
  Interventions: Drug: midazolam
- dexmedetomidine (Active Comparator): The patients will be given nebulized dexmedetomidine 2 μg/kg body weight 30 min before surgery.
  Interventions: Drug: dexmedetomidine

INTERVENTIONS:
Drug: fentanyl — nebulized fentanyl 2μg/kg body weigh
  Other Names: fentanyl,
  Arms: fentanyl
Drug: midazolam — nebulized midazolam 0.2 mg/kg body weight 30 min before surgery.
  Other Names: dormicum
  Arms: midazolam
Drug: dexmedetomidine — nebulized dexmedetomidine 2 μg/kg body weight 30 min before surgery.
  Other Names: precedex
  Arms: dexmedetomidine

SUMMARY:
* The preoperative time can be traumatic for young children undergoing surgery. Pediatric anesthesiologists act strongly to decrease distress for children in the operating room (OR) and to provide a smooth induction of anesthesia.
* Many drugs have been used as premedication to decrease anxiety , facilitate smooth induction and easy separation of children from their parents.
* This study was designed to evaluate and compare the effect and safety of nebulized either fentanyl, midazolam or nebulized dexmedetomidine as a sedative premedication prior to general anesthesia (GA) in outpatient pediatric dental surgeries.

DETAILED DESCRIPTION:
The preoperative time can be traumatic for young children undergoing surgery. Pediatric anesthesiologists act strongly to decrease distress for children in the operating room (OR) and to provide a smooth induction of anesthesia(1). Parentral separation and needle injection increase preoperative anxiety. Preoperative stress response stimulates the sympathetic, parasympathetic, and endocrine systems, leading to an increase in heart rate (HR), blood pressure, and cardiac excitability(2,3) . Dental procedures are assiociated by high rate of fear and anxiety in children (4).

Many drugs have been used as premedication to decrease anxiety , facilitate smooth induction and easy separation of children from their parents. The ideal premedication especially in children must be acceptable with rapid onset ,minimal side effects and with rapid postoperative recovery and return to alertness (5,6).

Fentanyl is a potent analgesic opioid with a rapid onset, and short duration of action (7). Midazolam is a short-acting benzodiazepine that has anxiolytic, amnestic, hypnotic, anticonvulsant and muscle relaxant actions (8,9). Dexmedetomidine is a selective α-2 adrenergic agonist that has both sedative and analgesic effects (10-12)

Preoperative sedation in children is usually administered via the rectal, oral sublingual, and intranasal routes with different degrees of patient acceptance.(13-18). Nebulized drug is an alternative method of sedation that is relatively easy to set up, without need for venipuncture, and is associated with high bioavailability of the drug (19,20).

This study was designed to evaluate and compare the effect and safety of nebulized either fentanyl, midazolam or nebulized dexmedetomidine as a sedative premedication prior to general anesthesia (GA) in outpatient pediatric dental surgeries. The primary end point is the time of sedation and level of sedation when the child is first seen in the operating room(OR) 30 minutes after using studied drugs, based on the Modified Observer's Assessment of Alertness/Sedation Scale(19). The secondary end points are parentral separation, tolerance to mask induction, reaction to intravenous cannulation, hemodynamic changes( systolic blood pressure, diastolic blood pressure and heart rate), sedation at emergence and wake-up behavior.

ELIGIBILITY:
Inclusion Criteria:

* Parent acceptance.Children 2-6 years old of either sex.12-18 kg body weight. american society of anesthesiologist I-II.outpatients dental surgeries under general anesthesia.

Exclusion Criteria:

Difficult airway .central nervous system dysfunction.Advanced Cardiovascular ,liver, renal diseases. Allergy to the drugs under study. Patients with any intranasal pathology or congenital anomaly.Patient refusal to take the inhaled premeditation.

Ages: 2 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 39 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2021-01-20 (Actual); Study Completion 2021-04-20 (Actual)

PRIMARY OUTCOMES:
of onset of sedation | Baseline (before surgery)
  onset of sedation based on the Modified Observer's Assessment of Alertness/Sedation Scale 6Appears alert and awake, responds readily to name spoken in normal tone 5 Appears asleep but responds readily to name spoken in normal tone 4 Lethargic response to name spoken in normal tone 3 Responds only after name is called loudly or repeatedly 2 Responds only after mild prodding or shaking
  1 Does not respond to mild prodding or shaking 0 Does not respond to noxious stimulus

SECONDARY OUTCOMES:
Heart rate | Baseline (before surgery) and intraoperative
  hemodynamic changes
systolic and diastolic blood pressure | Baseline (before surgery) and intraoperative
  hemodynamic changes

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine,Zagazig University, Zagazig, Zagazig, Elsharkia,egypt, Egypt

IPD SHARING:
Plan to Share IPD: Yes
planned after completion of the study and publication
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: planned after completion of the study and publication
Access Criteria: contact after pricipal investigator